CLINICAL TRIAL: NCT03347877
Title: Clinical Study of Autologous Osteo-periosteal Cylinder Graft Transplantation for Hepple V Osteochondral Lesions of the Talus
Brief Title: Autologous Osteo-periosteal Cylinder Graft Transplantation for Hepple V Osteochondral Lesions of the Talus
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Principal Investigator, Guo Qinwei, Principal Investigator, Clinical Associate Professor and Chief Orthopedist of Orthopedic Sports Medicine, Peking University Third Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PKU-GUO-01
Record Dates: First submitted 2017-11-15; First posted 2017-11-20 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-06

CONDITIONS: Osteochondral; Defect
Keywords: autologous osteo-periosteal cylinder graft; autologous osteochondral graft; randomized controlled trial; Hepple V osteochondral lesions of the talus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- autologous bone-periosteal graft (Experimental): The patients in experimental group will undergo the surgery of arthroscopic repair Hepple V osteochondral lesions of the talus with autologous osteo-periosteal cylinder graft transplantation.
  Interventions: Procedure: autologous osteo-periosteal cylinder graft transplantation; Device: autologous osteo-periosteal cylinder graft
- autologous osteochondral graft (Active Comparator): The patients in control group will undergo the surgery of arthroscopic repair Hepple V osteochondral lesions of the talus with autologous osteochondral graft transplantation.
  Interventions: Procedure: autologous osteochondral graft transplantation

INTERVENTIONS:
Procedure: autologous osteo-periosteal cylinder graft transplantation — Autologous osteo-periosteal cylinder graft transplantation is a novel treatment for Hepple V osteochondral lesions of the talus.
  Arms: autologous bone-periosteal graft
Procedure: autologous osteochondral graft transplantation — Autologous osteochondral graft transplantation is the most common treatment for Hepple V osteochondral lesions of the talus.
  Arms: autologous osteochondral graft
Device: autologous osteo-periosteal cylinder graft — Autologous osteo-periosteal cylinder graft is taken from ilium.
  Arms: autologous bone-periosteal graft

SUMMARY:
The trial evaluates the clinical efficacy and safety of autologous osteo-periosteal cylinder graft transplantation for Hepple V osteochondral lesions of the talus. Half of participants will receive autologous osteo-periosteal cylinder graft transplantation, while the other will receive osteochondral graft transplantation as a control group.

DETAILED DESCRIPTION:
Autologous osteo-periosteal cylinder graft surface is a periosteal structure, with the ability of repairment to cartilage, periosteum is closely connected to the cortical bone, then the deep loose cancellous bone.The objective of the study is to evaluate the clinical efficacy of autologous osteo-periosteal cylinder graft transplantation for Hepple V osteochondral lesions of the talus by randomized controlled trial. 70 patients with clinically diagnosed Hepple V talus osteochondral lesions according to 1: 1 were divided into experimental group and control group. The experimental group will be treated with autologous osteo-periosteal cylinder graft transplantation under arthroscopy. The control group will be treated with autologous osteochondral graft under arthroscopy. The patients will be treated by the same surgeon in this study group. Postoperative MRI MOCART evaluation, clinical AOFAS score, VAS score, Tegner score, and the secondary arthroscopy ICRS score will be selected as the measures of outcome. The incidence of adverse events will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* 18-50 years old, male or female
* Chronic pain in the ankle, confirmed by ankle joint MRI as Hepple V osteo-chondral lesions of the talus
* Using rest/external use/oral non-steroidal anti-inflammatory drugs and other conservative treatment for more than 3 months ineffective
* Patients voluntarily participated in clinical trials, signed informed consent, with clinical follow-up

Exclusion Criteria:

* In the last 6 months patients participated in other drug or medical device clinical trials
* Line of force in ankle is not correct (varus or valgus> 5 degrees)
* Grade III ankle collateral ligament injury
* Chronic specific synovitis (rheumatoid, pigmented villonodular synovitis, etc.)
* Joint fibrosis, ankylosis, activity was significantly limited
* Moderate and severe osteoarthritis
* There are MRI contraindications
* Hemophilia patients
* The general condition of patients can not tolerate surgery
* Pregnant or planned pregnant women and lactating women
* Abnormal mental capacity without autonomy
* Other conditions in which the doctor can not decide to participate in the trial

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
American Orthopaedic Foot & Ankle Society(AOFAS) ankle-hindfoot score | 4 years
  American Orthopaedic Foot & Ankle Society(AOFAS) ankle-hindfoot score. The higher score represent the better outcome.

SECONDARY OUTCOMES:
International Cartilage Repair Society(ICRS) score | 4 years
  International Cartilage Repair Society(ICRS) score. The higher score represent the better outcome.
Magnetic Resonance Observation of cartilage repair tissue(MOCART) score | 4 years
  Magnetic Resonance Observation of cartilage repair tissue(MOCART) score. The higher score represent the better outcome.
Tegner activity level score | 4 years
  The highest level of activity that you participated in before your injury and the highest level you are able to participate in currently. The higher values represent a better outcome.
Visual analogue scale | 4 years
  The visual analogue scale or visual analog scale (VAS) is a psychometric response scale which can be used in questionnaires. It is a measurement instrument for subjective characteristics or attitudes that cannot be directly measured. When responding to a VAS item, respondents specify their level of agreement to a statement by indicating a position along a continuous line between two end-points. From 0 to 10, no pain 0, worst pain imaginable 10. The higher values represent a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Qinwei Guo, Principal Investigator — Peking University Third Hospital
Locations (1):
- Institute of Sports Medicine, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yang S, Hu F, Shao Q, Zhang Z, Liu X, Jiang Y, Jiang D, Xie X, Jiao C, Hu Y, Shi W, Guo Q. Autologous Osteoperiosteal Transplantation Versus Autologous Osteochondral Transplantation for Large Cystic Osteochondral Lesions of the Medial Talus: 2-Year Results From a Prospective Randomized Controlled Trial. Am J Sports Med. 2025 Sep;53(11):2642-2651. doi: 10.1177/03635465251361505. Epub 2025 Aug 19. PMID 40828751
- [Derived] Deng E, Shi W, Jiang Y, Guo Q. Comparison of autologous osteoperiosteal cylinder and osteochondral graft transplantation in the treatment of large cystic osteochondral lesions of the talus (OLTs): a protocol for a non-inferiority randomised controlled trial. BMJ Open. 2020 Feb 9;10(2):e033850. doi: 10.1136/bmjopen-2019-033850. PMID 32041859